CLINICAL TRIAL: NCT06915389
Title: Comprehensive Plasma Metabolomic and Lipidomic Profiling for Predictive Modeling and Biomarker Discovery of Immune-Related Adverse Events in PD-1/PD-L1 Inhibitor-Treated Gastric Cancer Patients: A Prospective Cohort Study
Brief Title: Metabolomic and Lipidomic Analysis Predicts Immunotherapy-related Adverse Events in Gastric Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Qinghai Red Cross Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-02
Record Dates: First submitted 2025-02-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Immunotherapy; Adverse Event; Metabonomics; Lipidomics
Keywords: Immune-related adverse events (irAEs); PD-1/PD-L1 inhibitors; Gastric cancer; Biomarkers; Metabolic; Lipidomic
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immune-related adverse events（irAEs）group: Integrated metabolomic and lipidomic profiling was conducted to delineate the differential metabolic signatures and lipidomic alterations prior to PD-1/PD-L1 inhibitor therapy initiation and throughout the progression of immune-related adverse events (irAEs)
- Non-Immune-related adverse events (Non-irAEs) group: Integrated metabolomic and lipidomic profiling was conducted to delineate the differential metabolic signatures and lipidomic alterations prior to PD-1/PD-L1 inhibitor therapy initiation and throughout the progression of immune-related adverse events (irAEs)

SUMMARY:
This study comprehensively examines metabolic and lipidomic dynamics in gastric cancer patients initiating PD-1/PD-L1 inhibitor therapy, employing a longitudinal design with pre- and post-treatment patients. The primary objectives include identifying irAE-associated metabolic and lipid biomarkers, developing predictive risk models, and evaluating the prognostic value of these molecular profiles. The findings are expected to contribute significantly to personalized treatment strategies and improved clinical decision-making in immunooncology.

DETAILED DESCRIPTION:
This study is designed as a prospective clinical trial employing advanced metabolomics and lipidomics methodologies to comprehensively analyze alterations in metabolites and lipid molecules within plasma samples. The primary objective is to investigate the differential profiles between gastric cancer patients who induce immune-related adverse events (irAEs) and who not, following Programmed Cell Death Protein 1/Programmed Death-Ligand 1 inhibitor(PD-1/PD-L1 inhibitor) therapy. Through this approach, the investigators aim to establish predictive biomarkers for irAEs occurrence and subsequently develop a robust prognostic model to enhance clinical management and therapeutic outcomes. Patients who meet the inclusion and exclusion criteria will be formally enrolled after screening and signing an informed consent form. Patients pathologically confirmed of gastric cancer who received anti-PD-1/anti-PD-L1 blockade therapy alone or with combined with chemotherapy. Baseline plasma samples were collected before immune checkpoint inhibitors(ICIs) treatment for all patients. Patients with irAEs collected plasma samples at the onset of irAEs, and patients without irAEs collected samples according to the treatment cycles to onset of irAEs patients. Patients with irAEs and without irAEs were matched by 1:1 or 1:2 for consideration of age, sex and stage to confirm the sample of which cycle should be chosen for patients without irAEs. Comprehensive metabolomics and lipidomics analyses were performed on the collected plasma samples,Differential metabolites and lipid molecules related to immune-related adverse events were screened out.By leveraging the identified key metabolites and lipid molecules, a robust predictive model has been developed to evaluate the risk of immune-related adverse events in patients. Comprehensive data on quality-of-life metrics and adverse event severity grading were systematically collected for patients experiencing immune-related adverse events. Extended analyses were carried out to evaluate potential links between the identified metabolic/lipidomic signatures and long-term patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years

  * ECOG PS 0-2

    * Gastric cancer diagnosed by histology or cytology

      * Untreatment with PD-1/PD-L1 inhibitors

        * Expected survival≥3 months

          * Exhibits a favorable adherence to treatment and follow-up,demonstrates compliance with the research protocol, and willingly signs the informed consent form.

Exclusion Criteria:

* Unable to obtain an organization or due to insufficient organizational material, unable to diagnose gastric cancer

  * Refusal to receive PD-1/PD-L1 inhibitor treatment

    * Baseline (before immunotherapy) plasma samples are unavailable

      * Combined with autoimmune diseases

        * Baseline (before immunotherapy) there are severe diseases in the heart, lungs, thyroid gland and other organs

          * Baseline (before immunotherapy) there are severe abnormalities in liver and kidney functions, pancreatic enzymes and other indicators

            ⑦ Researchers posit that any condition deemed potentially harmful to the subjects or that might prevent subjects from meeting or adhering to the research requirements shall not be permissible for inclusion in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the research subjects were patients with gastric cancer who were aged ≥ 18 years, had ECOG score ranging from 0 to 2, were confirmed by pathology, and received either anti-PD-L1/anti-PD-1 monotherapy or combination chemotherapy, with an expected survival period of ≥ 3 months
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of immune-related adverse events | 1 year
  * For gastric cancer patients receiving immunotherapy for the first time, immune-related adverse events should be monitored during treatment, with a follow-up period of 1 year.
    * The immune checkpoint inhibitors include pembrolizumab, nivolumab, sintilimab, tislelizumab, sugemalimab and camrelizumab.
      * NCCN Guidelines for Management of Immunotherapy-Related Toxicity are adopted as the gold standard for assessing immune-related adverse events.
        * The severity of immune-related adverse events was evaluated based on the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Changes in Plasma Metabolite Levels | 1 year
  * A comprehensive metabolomic profiling of plasma in treatment-naïve gastric cancer patients undergoing immunotherapy: Investigating metabolic disparities between responders with immune-related adverse events and those without.
    * The measurement methods include gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS).
      * The measured metabolites include amino acids, fatty acids, glucose, lactate, nucleotides, organic acids, vitamins and small-molecule metabolites.
        * All metabolomic markers in plasma will be reported as relative quantitative values in arbitrary units.
          * Baseline plasma samples were collected from all patients prior to immunotherapy, and follow-up samples were obtained every 2 treatment cycles until 1 year after treatment initiation.
Changes in Plasma Lipid Levels | 1 year
  * Comprehensive lipidomic profiling of plasma from gastric cancer patients undergoing initial immunotherapy was performed to investigate differential plasma lipid signatures between those who developed immune-related adverse events and those who did not.
    * The measurement methods include gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS).
      * The measured lipids include triglycerides, cholesterol, phospholipids, fatty acids, ceramides, steroids, fatty acid derivatives, and other sphingolipids.
        * All plasma lipidomic markers will be reported as relative quantitative values in arbitrary units.
          * Baseline plasma samples were collected from all patients prior to immunotherapy, with subsequent samples obtained every 2 treatment cycles until 1 year of therapy.

SECONDARY OUTCOMES:
Develop a predictive model for immune-related adverse events | 2 years
  * This predictive model incorporates input variables including lipid molecules, metabolites, and baseline clinical characteristics of patients, with the output being an adverse event risk score (low, intermediate, or high risk).
    * Employing machine learning algorithms (e.g., logistic regression, random forests, support vector machines) to construct predictive models.
      * The clinical characteristics include age (reported in years), height and weight (reported as BMI in kg/m²), gender (recorded as male or female), tumor stage (classified by TNM staging system).
        * The measured metabolites include amino acids, fatty acids, glucose, lactate, nucleotides, organic acids, vitamins and small-molecule metabolites.
          * The measured lipids include triglycerides, cholesterol, phospholipids, fatty acids, ceramides, steroids, fatty acid derivatives, and other sphingolipids.
            * All metabolomic and lipidomics markers in plasma will be reported as relative quantitative values in arbitrary units.
Investigating the correlation between metabolomic and lipidomic profiles and patient outcomes to inform evidence-based clinical decision-making. | 2 years
  Using survival analysis (e.g., Kaplan-Meier curves, Cox regression models) to assess the association between Immune-related adverse events and patient survival rates or recurrence rates

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai Red Cross Hospital, Xining, Qinghai, China